CLINICAL TRIAL: NCT07286526
Title: Comparison of Bolus and Continuous Hydration Regimens for the Prevention of Contrast-Associated Acute Kidney Injury in the Emergency Department: A Randomized Controlled Non-Inferiority Trial
Brief Title: Comparison of Bolus and Continuous Hydration Regimens for the Prevention of Contrast-Associated Acute Kidney Injury in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yunus Emre Gemici (Other Government)
Responsible Party: Sponsor-Investigator, Yunus Emre Gemici, MD, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-66291034-202.3.02-4819
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury Following Administration of Contrast Media
Keywords: non-inferiorty; randomized controlled trial; contrast associated acute kidney injury; contrast agents; hydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus hydration therapy (Experimental): In the Bolus hydration therapy group, 500 ml of 0.9% saline treatment was started half an hour before the procedure and after the procedure, 1000 ml of 0.9% saline treatment was continued at a rate of 500 ml/h to be completed in 2 hours. A total of 1500 ml 0.9% saline hydration therapy was administered over 2.5 hours. According to the literature, individuals with an ejection fraction of less than 40% got a half-dose hydration protocol. In the bolus hydration group, 250 ml of treatment was administered half an hour before the procedure, and hydration was continued at a rate of 250 ml/h for 2 hours after the procedure.
  Interventions: Drug: Bolus hydration therapy
- Continuous hydration therapy (Active Comparator): In the Continuous hydration therapy group, saline treatment started 2 hours before the intravenous (IV) contrast agent application at a rate of 150 ml/h, and hydration was applied for 8 more hours after the procedure at the same rate. A total of 1500 ml 0.9% saline hydration therapy was administered over 10 hours. According to the literature, individuals with an ejection fraction of less than 40% got a half-dose hydration protocol. In the continuous hydration group, 75 ml/h of hydration was administered for 2 hours before the procedure and for 8 hours after the procedure.
  Interventions: Drug: Continuous hydration therapy

INTERVENTIONS:
Drug: Bolus hydration therapy — In the Bolus hydration therapy group, 500 ml of 0.9% saline treatment was started half an hour before the procedure and after the procedure, 1000 ml of 0.9% saline treatment was continued at a rate of 500 ml/h to be completed in 2 hours. A total of 1500 ml 0.9% saline hydration therapy was administered over 2.5 hours. According to the literature, individuals with an ejection fraction of less than 40% got a half-dose hydration protocol. In the bolus hydration group, 250 ml of treatment was administered half an hour before the procedure, and hydration was continued at a rate of 250 ml/h for 2 hours after the procedure.
  Arms: Bolus hydration therapy
Drug: Continuous hydration therapy — In the Continuous hydration therapy group, saline treatment started 2 hours before the intravenous (IV) contrast agent application at a rate of 150 ml/h, and hydration was applied for 8 more hours after the procedure at the same rate. A total of 1500 ml 0.9% saline hydration therapy was administered over 10 hours. According to the literature, individuals with an ejection fraction of less than 40% got a half-dose hydration protocol. In the continuous hydration group, 75 ml/h of hydration was administered for 2 hours before the procedure and for 8 hours after the procedure.
  Arms: Continuous hydration therapy

SUMMARY:
A single-center, prospective, open-label, non-inferiority randomized controlled clinical trial was conducted at the ED of a tertiary hospital. The ED staff consisted of a mix of emergency medicine specialists, emergency medicine residents, and general practitioners.

Between August 10, 2024, and March 26, 2025, patients aged 18 and over who presented to the ED with creatinine levels above the reference range (1.2 mg/dl in men and 1.1 mg/dl in women) and underwent contrast-enhanced tomography were deemed eligible for inclusion in the study.

Eligible patients were randomly allocated in a 1:1 ratio to receive either bolus hydration or continuous hydration therapy. Permuted block randomization was employed at each participating site to distribute patients, stratified by age groups (18-44, 45-59, 60-74, and 75 years and older) and gender. This study did not use blinding. Both the implementers of the intervention and the researchers evaluating the outcome measures are aware of the intervention groups.

After the patients were divided into two groups, one group received bolus hydration therapy while the other group received continuous hydration therapy.

According to the literature, individuals with an ejection fraction of less than 40% got a half-dose hydration protocol.

The IV contrast agent used in the study was iohexol, which belongs to the non-ionic low osmolar contrast agent group. 300 mgI/ml 100 ml solutions were used, and the dose was adjusted between 80 and 100 ml depending on the imaging and the patient. In the majority of patients, 100 ml of contrast was administered, with an average of 98 ml of solution given in the bolus hydration group and an average of 96 ml of solution given in the continuous hydration group.

Patients were given control forms to provide follow-up blood samples 48-72 hours later and were asked to present to the ED with the form on the specified date. To inquire about the development of dialysis needs and mortality status, patients were contacted 30 days later to gather information.

ELIGIBILITY:
Inclusion Criteria:

* Presented to the Emergency Department creatinine levels above the reference range (1.2 mg/dl in men and 1.1 mg/dl in women)
* Underwent contrast-enhanced tomography

Exclusion Criteria:

* Pregnancy
* Known allergy history to contrast agents
* Exposure to contrast agents within the last 72 hours
* Being on dialysis due to end-stage kidney disease
* Presenting with decompensated heart failure
* Patients who were unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-03-29 (Actual); Study Completion 2025-04-26 (Actual)

PRIMARY OUTCOMES:
Rate of Participants Who Developed Contrast-Associated Acute Kidney Injury (CA-AKI) | From enrollment to the end of treatment at 1 week
  The primary outcome of our study was the development of CA-AKI, defined as an increase in serum creatinine value by ≥25% compared to baseline or an absolute increase in serum creatinine value by ≥0.5 mg/dL within 48-72 hours after contrast administration.

SECONDARY OUTCOMES:
Rate of Participants Who Required Dialysis | From enrollment to the end of treatment at 1 month
  Patients were contacted by phone 1 month after the procedure and asked about the development of dialysis needs within that 1-month period.
All-Cause Mortality Rate | From enrollment to the end of treatment at 1 month
  Patients were contacted by phone 1 month after the procedure and asked about the all-cause Mortality within that 1-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Çalık, MD, Assoc. Prof., Study Director — Department of Emergency Medicine Gaziosmanpaşa Training and Research Hospital, İstanbul, Türkiye
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves single-center clinical data without a dedicated data-sharing infrastructure, and sharing these data may pose risks to participant privacy despite de-identification efforts.

REFERENCES:
- [Background] Katzberg RW, Newhouse JH. Intravenous contrast medium-induced nephrotoxicity: is the medical risk really as great as we have come to believe? Radiology. 2010 Jul;256(1):21-8. doi: 10.1148/radiol.10092000. No abstract available. PMID 20574082
- [Background] James MT, Samuel SM, Manning MA, Tonelli M, Ghali WA, Faris P, Knudtson ML, Pannu N, Hemmelgarn BR. Contrast-induced acute kidney injury and risk of adverse clinical outcomes after coronary angiography: a systematic review and meta-analysis. Circ Cardiovasc Interv. 2013 Feb;6(1):37-43. doi: 10.1161/CIRCINTERVENTIONS.112.974493. Epub 2013 Jan 15. PMID 23322741
- [Background] Cho E, Ko GJ. The Pathophysiology and the Management of Radiocontrast-Induced Nephropathy. Diagnostics (Basel). 2022 Jan 12;12(1):180. doi: 10.3390/diagnostics12010180. PMID 35054347
- [Background] Ehmann MR, Klein EY, Zhao X, Mitchell J, Menez S, Smith A, Levin S, Hinson JS. Epidemiology and Clinical Outcomes of Community-Acquired Acute Kidney Injury in the Emergency Department: A Multisite Retrospective Cohort Study. Am J Kidney Dis. 2024 Jun;83(6):762-771.e1. doi: 10.1053/j.ajkd.2023.10.009. Epub 2023 Dec 10. PMID 38072210
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. Circulation. 2011 Dec 6;124(23):e574-651. doi: 10.1161/CIR.0b013e31823ba622. Epub 2011 Nov 7. No abstract available. PMID 22064601
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Blackwelder WC. "Proving the null hypothesis" in clinical trials. Control Clin Trials. 1982 Dec;3(4):345-53. doi: 10.1016/0197-2456(82)90024-1. PMID 7160191
- [Background] Sebastia C, Paez-Carpio A, Guillen E, Pano B, Garcia-Cinca D, Poch E, Oleaga L, Nicolau C. Oral hydration compared to intravenous hydration in the prevention of post-contrast acute kidney injury in patients with chronic kidney disease stage IIIb: A phase III non-inferiority study (NICIR study). Eur J Radiol. 2021 Mar;136:109509. doi: 10.1016/j.ejrad.2020.109509. Epub 2021 Jan 14. PMID 33516141
- [Background] Lombardi M, Molisana M, Genovesi E, De Innocentiis C, Limbruno U, Misuraca L, Moretti L, Di Vito L, Renda G, Zimarino M, Di Nicola M, De Caterina R. Urine alkalinisation to prevent contrast-induced acute kidney injury: the prospective, randomised, controlled, open-label TEATE trial. EuroIntervention. 2022 Sep 20;18(7):562-573. doi: 10.4244/EIJ-D-22-00010. PMID 35620986
- [Background] Ravn EJ, Hasific S, Thomassen M, Hjortebjerg R, Bach Laursen K, Diederichsen A, Bistrup C, Ovrehus KA. Intravenous versus oral hydration to reduce the risk of postcontrast acute kidney injury after intravenous contrast-enhanced CT in patients with severe chronic kidney disease (ENRICH): a study protocol for a single-centre, parallel-group, open-labelled non-inferiority randomised controlled trial in Denmark. BMJ Open. 2023 Sep 12;13(9):e074057. doi: 10.1136/bmjopen-2023-074057. PMID 37699636
- [Background] Somkereki C, Palfi R, Scridon A. Prevention of contrast-associated acute kidney injury in an era of increasingly complex interventional procedures. Front Med (Lausanne). 2024 Jan 9;10:1180861. doi: 10.3389/fmed.2023.1180861. eCollection 2023. PMID 38264052
- [Background] Section 4: Contrast-induced AKI. Kidney Int Suppl (2011). 2012 Mar;2(1):69-88. doi: 10.1038/kisup.2011.34. No abstract available. PMID 25018920
- [Background] Li Y, Wang J. Contrast-induced acute kidney injury: a review of definition, pathogenesis, risk factors, prevention and treatment. BMC Nephrol. 2024 Apr 22;25(1):140. doi: 10.1186/s12882-024-03570-6. PMID 38649939
- [Background] Arslan S, Yildiz A, Dalgic Y, Batit S, Kilicarslan O, Ser OS, Dalgic SN, Kocas C, Abaci O. Avoiding the emergence of contrast-induced acute kidney injury in acute coronary syndrome: routine hydration treatment. Coron Artery Dis. 2021 Aug 1;32(5):397-402. doi: 10.1097/MCA.0000000000000966. PMID 33060531
- [Background] Liu Y, Tan N, Huo Y, Chen S, Liu J, Chen YD, Wu K, Wu G, Chen K, Ye J, Liang Y, Feng X, Dong S, Wu Q, Ye X, Zeng H, Zhang M, Dai M, Duan CY, Sun G, He Y, Song F, Guo Z, Chen PY, Ge J, Xian Y, Chen J. Hydration for prevention of kidney injury after primary coronary intervention for acute myocardial infarction: a randomised clinical trial. Heart. 2022 May 25;108(12):948-955. doi: 10.1136/heartjnl-2021-319716. PMID 34509996
- [Background] Liu Y, Tan N, Huo Y, Chen SQ, Liu J, Wang Y, Li L, Tao JH, Su X, Zhang L, Li QX, Zhang JY, Guo YS, Du ZM, Zhou YP, Fang ZF, Xu GM, Liang Y, Tao L, Chen H, Ji Z, Han B, Chen PY, Ge JB, Han YL, Chen JY. Simplified Rapid Hydration Prevents Contrast-Associated Acute Kidney Injury Among CKD Patients Undergoing Coronary Angiography. JACC Cardiovasc Interv. 2023 Jun 26;16(12):1503-1513. doi: 10.1016/j.jcin.2023.03.025. PMID 37380233
- [Background] Chen F, Lu J, Yang X, Liu D, Wang Q, Geng X, Xiao B, Zhang J, Liu F, Gu G, Cui W. Different hydration methods for the prevention of contrast-induced nephropathy in patients with elective percutaneous coronary intervention: a retrospective study. BMC Cardiovasc Disord. 2023 Jun 24;23(1):323. doi: 10.1186/s12872-023-03358-w. PMID 37355592
- [Background] Hoste EAJ, Kellum JA, Selby NM, Zarbock A, Palevsky PM, Bagshaw SM, Goldstein SL, Cerda J, Chawla LS. Global epidemiology and outcomes of acute kidney injury. Nat Rev Nephrol. 2018 Oct;14(10):607-625. doi: 10.1038/s41581-018-0052-0. PMID 30135570
- [Background] Batte A, Shahrin L, Claure-Del Granado R, Luyckx VA, Conroy AL. Infections and Acute Kidney Injury: A Global Perspective. Semin Nephrol. 2023 Sep;43(5):151466. doi: 10.1016/j.semnephrol.2023.151466. Epub 2023 Dec 28. PMID 38158245
- [Background] Kellum JA, Romagnani P, Ashuntantang G, Ronco C, Zarbock A, Anders HJ. Acute kidney injury. Nat Rev Dis Primers. 2021 Jul 15;7(1):52. doi: 10.1038/s41572-021-00284-z. PMID 34267223
- [Background] Section 1: Introduction and Methodology. Kidney Int Suppl (2011). 2012 Mar;2(1):13-18. doi: 10.1038/kisup.2011.31. No abstract available. PMID 25018917
- See also: Related Info — https://www.sealedenvelope.com/power/binary-noninferior/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT07286526/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT07286526/ICF_001.pdf